CLINICAL TRIAL: NCT00175890
Title: A Double-Blind, Randomized, Multicenter, Placebo-controlled, In-Patient, Maximum 34 Day Study of Levetiracetam Oral Solution (20-50 mg/kg/Day) as Adjunctive Treatment of Refractory Partial Onset Seizures in Pediatric Epileptic Subjects Ranging in Age From 1 Month to Less Than 4 Years of Age
Brief Title: A Placebo-controlled Study of Levetiracetam In Children (1mo to 4yrs of Age) With Partial Onset Seizures.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01009; 2004-000199-14 (EudraCT Number)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Epilepsy, Partial
Keywords: Partial Onset Seizure; levetiracetam; Video Electroencephalogram; Keppra
MeSH Terms: conditions — Epilepsies, Partial | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matching oral solution to Levetiracetam b.i.d. (twice a day) for a maximum treatment duration of 20 days.
  Interventions: Other: Placebo
- Levetiractem (Experimental): 10 % oral solution Levetiracetam b.i.d. (twice a day) for a maximum treatment duration of 20 days.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Dosing was stratified by age. A dose of 20 mg/kg/day titrating to 40 mg/kg/day for children one month to less than six months old and a dose of 25 mg/kg/day titrating to 50 mg/kg/day for children 6 month to less than 4 years old, was used in this study. The total daily dose was administered b.i.d.
  Other Names: Keppra
  Arms: Levetiractem
Other: Placebo — Placebo solution, which is indistinguishable from the Levetiracetam oral solution.
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of levetiracetam used as adjunctive treatment in pediatric subjects age 1 month to less than 4 years with partial onset seizures. Subjects will be evaluated with 48 hour inpatient video electroencephalograms (a selection and an evaluation). Other neuropsychological clinical assessments will be performed during the 34 day length of the study.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients from 1 month to less than 4 years of age
* Pediatric patients diagnosed with refractory partial onset seizures, on a stable regimen of one to two other anti-epileptic drugs and at least 2 partial onset seizures per week in the two weeks prior to screening
* Patients must have two partial onset seizures (with corresponding clinical event) during the 48-hour video EEG at screening

Exclusion Criteria:

* A ketogenic diet
* Previous exposure to levetiracetam
* Seizures too close together to count accurately
* Treatable seizure etiology
* Current diagnosis of Lennox-Gastaut Syndrome or epilepsy secondary to a progressing cerebral disease
* Diagnosis of a terminal illness

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2004-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Responder Rate for total partial onset seizures as computed from the 48-hour Evaluation video-EEG (post-baseline) and the 48-hour Selection video-EEG (baseline) | 48-hours in Evaluation Period and 48-hours in Selection Period
  Responder Rate is defined as the number of subjects with a ≥ 50 % reduction from baseline in their Average Daily Frequency (ADF) for partial onset seizures divided by the total number of subjects. If a subject had < 24 hours of usable Evaluation video-EEG time (including zero time available) and withdrawal from the study with reasons linked to lack or loss of efficacy, the subject was counted as a non-responder.

SECONDARY OUTCOMES:
Responder rate for total seizures (all types) as computed from the 48-hour Evaluation video-EEG (post-baseline) and the 48-hour Selection video-EEG (baseline) | 48-hours in Evaluation Period and 48-hours in Selection Period
  Responder Rate is defined as the number of subjects with a ≥ 50 % reduction from baseline in their Average Daily Frequency (ADF) for all seizure types divided by the total number of subjects. Subjects who withdrew or dropped out before the first 24 hours Evaluation video-EEG with reasons linked to lack of efficacy were considered as non-responders. All (total) seizures were defined as the total of Type I (partial onset) + Type II (Primary generalized) + Type III (unclassified epileptic).
Percent reduction in Average Daily Frequency (ADF) of partial onset seizures recorded on the 48-hour Evaluation video-EEG compared to those recorded on the 48-hour Selection video-EEG | 48-hours in Evaluation Period and 48-hours in Selection Period
  A positive value in Percent reduction from Selection Period to Evaluation Period indicates an improvement.
Percent reduction in Average Daily Frequency (ADF) of total seizures (all types) recorded on the 48-hour Evaluation video-EEG compared to those recorded on the 48-hour Selection video-EEG | 48-hours in Evaluation Period and 48-hours in Selection Period
  A positive value in Percent reduction from Selection Period to Evaluation Period indicates an improvement. All (total) seizures were defined as the total of Type I (partial onset) + Type II (Primary generalized) + Type III (unclassified epileptic).
Absolute reduction in Average Daily Frequency (ADF) of partial onset seizures recorded on the 48-hour Evaluation video-EEG compared to those recorded on the 48-hour Selection video-EEG | 48-hours in Evaluation Period and 48-hours in Selection Period
  A positive value in Absolute reduction from Selection Period to Evaluation Period indicates an improvement.
Absolute reduction in Average Daily Frequency (ADF) of total seizures (all types) recorded on the 48-hour Evaluation video-EEG compared to those recorded on the 48-hour Selection video-EEG | 48-hours in Evaluation Period and 48-hours in Selection Period
  A positive value in Absolute reduction from Selection Period to Evaluation Period indicates an improvement. All (total) seizures were defined as the total of Type I (partial onset) + Type II (Primary generalized) + Type III (unclassified epileptic).
Percent reduction in Average Daily Frequency (ADF) of electro-clinical partial onset seizures recorded on the 48-hour Evaluation video-EEG compared to those recorded on the 48-hour Selection video-EEG for children 1 month to less than 6 months old | 48-hours in Evaluation Period and 48-hours in Selection Period
  A positive value in Percent reduction from Selection Period to Evaluation Period indicates an improvement. For children 1 month to less than 6 months old, partial onset seizure counts were based on electroclinical seizures plus electrographic seizures.
Percentage of drop-outs for any reasons during the study | During the study (up to 20 days)
Percentage of drop-outs due to lack of efficacy during the study | During the study (up to 20 days)
Percentage of drop-outs before 24 hours of Evaluation video-EEG for reasons other than lack or loss of efficacy | During the study (up to 20 days)
Time to Exit (TTE) during the Evaluation Period | During Evaluation Period (Day 1 to Day 6)
  For early termination subjects in the Evaluation period the TTE is the time to discontinuing the study for any reason. TTE was defined as the day of study discontinuation - the day of randomization + 1. For completed subjects, the TTE was censored on Day 6.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (86):
- United States (42):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Gainesville, Florida
  - Loxahatchee Groves, Florida
  - Miami, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - Saint Paul, Minnesota
  - Lebanon, New Hampshire
  - Cherry Hill, New Jersey
  - Edison, New Jersey
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Danville, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Spartanburg, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Argentina (3):
  - Buenos Aires
  - Mendoza
  - Pilar Buenos Aires
- Belgium (2):
  - Brussels
  - Leuven
- Brazil (6):
  - Campinas
  - Curitiba
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - São Paulo
- Canada (6):
  - Vancouver, British Columbia
  - Winnepeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - London, Ontario
  - Scarborough Village, Ontario
  - Saskatoon, Saskatchewan
- Czechia (2):
  - Brno
  - Prague
- France (4):
  - Lille
  - Paris
  - Rouen
  - Strasbourg
- Germany (6):
  - Kehl, Kork
  - Berlin
  - Erlangen
  - Heidelberg
  - Jena
  - Kiel
- Budapest, Hungary
- Italy (4):
  - Calambrone
  - Genoa
  - Milan
  - Roma
- Mexico City, Mexico
- Gdansk, Poland
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Târgu Mureş
- Russia (3):
  - Kalingrad
  - Moscow
  - Saint Petersburg
- United Kingdom (2):
  - Glasgow
  - London

REFERENCES:
- [Result] Pina-Garza JE, Nordli DR Jr, Rating D, Yang H, Schiemann-Delgado J, Duncan B; Levetiracetam N01009 Study Group. Adjunctive levetiracetam in infants and young children with refractory partial-onset seizures. Epilepsia. 2009 May;50(5):1141-9. doi: 10.1111/j.1528-1167.2008.01981.x. Epub 2009 Feb 21. PMID 19243423
- [Derived] Pina-Garza JE, Schiemann-Delgado J, Yang H, Duncan B, Hadac J, Hunter SJ. Adjunctive levetiracetam in patients aged 1 month to <4 years with partial-onset seizures: subpopulation analysis of a prospective, open-label extension study of up to 48 weeks. Clin Ther. 2010 Oct;32(11):1935-50. doi: 10.1016/j.clinthera.2010.09.017. PMID 21095488